CLINICAL TRIAL: NCT02486627
Title: A Phase 3, Randomized, Multicenter, Double-Blind Study to Evaluate the Efficacy and Safety of Plazomicin Compared With Meropenem Followed by Optional Oral Therapy for the Treatment of Complicated Urinary Tract Infection (cUTI), Including Acute Pyelonephritis (AP), in Adults
Brief Title: A Study of Plazomicin Compared With Meropenem for the Treatment of Complicated Urinary Tract Infection (cUTI) Including Acute Pyelonephritis (AP)
Acronym: EPIC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Achaogen, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACHN-490-009; 2015-001588-37 (EudraCT Number); U1111-1171-1554 (Other: WHO)
Record Dates: First submitted 2015-06-25; First posted 2015-07-01 (Estimated); Results first posted 2018-08-23 (Actual); Last update posted 2018-08-23 (Actual); Status verified 2018-07

CONDITIONS: Complicated Urinary Tract Infection; Acute Pyelonephritis
Keywords: cUTI; AP; ACHN-490; anti-infective; anti-bacterial; antibiotic; anti-microbial; UTI; bacterial infection; Gram-negative
MeSH Terms: conditions — Bacterial Infections | interventions — plazomicin; Meropenem; Levofloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Plazomicin (Experimental): Patients received 15 milligrams per kilogram (mg/kg) plazomicin as an intravenous (IV) infusion once daily followed by matching placebo infusions 8 and 16 hours later. After a minimum of 4 days of IV plazomicin, patients could switch to 250 or 500 mg oral levofloxacin for a total duration of 7 to 10 days (IV plus oral).
  Interventions: Drug: plazomicin; Drug: levofloxacin (oral)
- Meropenem (Active Comparator): Patients received 1.0 g meropenem as an IV infusion every 8 hours (q8h). After a minimum of 4 days of IV meropenem, patients could switch to 250 or 500 mg oral levofloxacin for a total duration of 7 to 10 days (IV plus oral).
  Interventions: Drug: meropenem; Drug: levofloxacin (oral)

INTERVENTIONS:
Drug: plazomicin
  Arms: Plazomicin
Drug: meropenem
  Arms: Meropenem
Drug: levofloxacin (oral)

SUMMARY:
This was a randomized, multicenter, multinational, double-blind study comparing the efficacy and safety of plazomicin compared with meropenem followed by optional oral (PO) therapy in the treatment of cUTI, including AP, in adults.

ELIGIBILITY:
Key Inclusion Criteria:

* Pyuria
* Have a pretreatment baseline urine culture obtained within 36 hours before the start of administration of the first dose of study drug
* Clinical signs and/or symptoms of acute pyelonephritis or complicated urinary tract infection
* Normal renal function or moderate renal impairment

Key Exclusion Criteria:

* Confirmed fungal urinary tract infection at the time of randomization
* Known urinary tract infection or colonization with Gram-positive pathogens
* Current cUTI or AP is known to be caused by a pathogen resistant to meropenem
* Female participants of childbearing potential if they are known to be pregnant or have a positive pregnancy test at screening, breastfeeding, or unable or unwilling to use a highly effective method of birth control during the study and for at least 30 days following the last dose of study medication
* Any rapidly progressing disease or immediately life-threatening illness
* Documented presence of immunodeficiency or an immunocompromised condition
* Documented or known history of otologic surgery or disease including use of hearing aid, head injury leading to otologic damage, Ménière's disease, tumor of the head, neck, or auditory system, perilymphatic fistula, or autoimmune disease of the inner ear, or family history of hearing loss (excluding age-related hearing loss [onset after age of 65 years])

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 609 (Actual)
Dates: Start 2016-01-11 (Actual); Primary Completion 2016-09-22 (Actual); Study Completion 2016-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E Connolly, MD, PhD, Study Director — Achaogen, Inc.

REFERENCES:
- [Derived] Wagenlehner FME, Cloutier DJ, Komirenko AS, Cebrik DS, Krause KM, Keepers TR, Connolly LE, Miller LG, Friedland I, Dwyer JP; EPIC Study Group. Once-Daily Plazomicin for Complicated Urinary Tract Infections. N Engl J Med. 2019 Feb 21;380(8):729-740. doi: 10.1056/NEJMoa1801467. PMID 30786187

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Plazomicin | Meropenem
Started | 306 | 303
Completed | 299 | 294
Not Completed | 7 | 9
Not completed — Death | 1 | 0
Not completed — Other Unspecified | 0 | 2
Not completed — Consent Withdrawn by Participant | 4 | 3
Not completed — Significant Participant Noncompliance | 1 | 1
Not completed — Lost to Follow-up | 1 | 3

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population includes all randomized patients.
Groups:
- Plazomicin: Patients received up to 15 mg/kg plazomicin as an IV infusion once daily followed by matching placebo infusions 8 and 16 hours later. After a minimum of 4 days of IV plazomicin, patients could switch to 250 or 500 mg oral levofloxacin for a total duration of 7 to 10 days (IV plus oral).
- Meropenem: Patients received 1.0 g meropenem as an IV infusion q8h. After a minimum of 4 days of IV meropenem, patients could switch to 250 or 500 mg oral levofloxacin for a total duration of 7 to 10 days (IV plus oral).
- Total: Total of all reporting groups
Arm/Group | Plazomicin | Meropenem | Total
Number analyzed (Participants) | 306 | 303 | 609
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.2 (18.29) | 59 (17.62) | 58.6 (17.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 171 | 149 | 320
  Male | 135 | 154 | 289
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 304 | 302 | 606
  Black or African American | 1 | 0 | 1
  Asian | 0 | 0 | 0
  American Indian or Native American | 0 | 0 | 0
  Native Hawaiin/Other Pacific Islander | 0 | 0 | 0
  Other Unspecified | 1 | 1 | 2
  Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients With Composite of Microbiological Eradication and Clinical Cure in the Microbiological Modified ITT (mMITT) Population at Day 5
Description: Microbiological eradication was defined as a urine culture that showed the pathogen found at baseline at ≥10^5 colony forming units per milliliter (CFU/mL) was reduced to <10^4 CFU/mL. Clinical Cure at Day 5: marked improvement evidenced by complete resolution or return to premorbid levels or reduction in severity of all core baseline symptoms with worsening of none, and no new symptoms developed. Failure: Lack of improvement in core baseline symptoms of cUTI or development of new core symptoms of cUTI; adverse event (AE) requiring the discontinuation of study drug and the patient required alternative non-study antibiotic therapy for the current cUTI. Indeterminate: Insufficient data are available to allow an evaluation of clinical outcome for any reason.
Time Frame: Day 5
Population: The mMITT Population consisted of all patients in the ITT Population who received any amount of study drug and had at least one qualified baseline pathogen from a study qualifying baseline urine culture against which meropenem and plazomicin have antibacterial activity.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin | Meropenem
Number analyzed (Participants) | 191 | 197
percentage of patients
  Composite Cure | 88 | 91.4
  Composite Failure | 10.5 | 7.6
  Indeterminate | 1.6 | 1
Statistical Analysis 1: Comparison: Plazomicin vs Meropenem; Test type: Non-Inferiority — 95% CIs for the difference in cure rates were calculated using the Newcombe method with continuity correction; Difference = -3.4, 95% CI 2-sided [-10 to 3.1]

2. Primary Outcome: Percentage of Patients With Composite of Microbiological Eradication and Clinical Cure in the mMITT Population at Test of Cure (TOC)
Description: Microbiological eradication was defined as a urine culture that showed the pathogen found at baseline at ≥10^5 CFU/mL was reduced to <10^4 CFU/mL. Clinical Cure at TOC Visit: the complete resolution or return to premorbid levels of core symptoms of cUTI and no new symptoms develop, and no use of non-study antibiotic therapy for the current cUTI. Failure: Persistence of one or more core symptom of infection or reappearance of or development of new core symptoms that require alternative non-study antibiotic therapy for the current cUTI. Indeterminate: Insufficient data are available to allow an evaluation of clinical outcome for any reason.
Time Frame: Day 17 TOC Visit
Population: as for outcome 1
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin | Meropenem
Number analyzed (Participants) | 191 | 197
percentage of patients
  Composite Cure | 81.7 | 70.1
  Composite Failure | 15.2 | 25.9
  Indeterminate | 3.1 | 4.1
Statistical Analysis 1: Comparison: Plazomicin vs Meropenem; Test type: Non-Inferiority — 95% CIs for the difference in cure rates were calculated using the Newcombe method with continuity correction; Difference = 11.6, 95% CI 2-sided [2.7 to 20.3]

3. Secondary Outcome: Percentage of Patients With Composite of Microbiological Eradication and Clinical Cure in the ME Population at Day 5
Description: Microbiological eradication: urine culture showed the pathogen found at baseline at ≥10^5 CFU/mL was reduced to <10^4 CFU/mL. Clinical Cure Day 5: Marked improvement defined as complete resolution or return to premorbid levels or reduction in severity of all core baseline symptoms with worsening of none, and no new symptoms develop. Failure Day 5: Lack of improvement in core baseline symptoms of cUTI or development of new core symptoms of cUTI; AE requiring the discontinuation of study drug and the patient required alternative non-study antibiotic therapy for the current cUTI.
Time Frame: Day 5
Population: The ME (Day 5) population consists of clinically evaluable patients with interpretable culture results at Day 5, defined as one that has clearly identified pathogen(s) or one where baseline pathogen(s) could be excluded.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin | Meropenem
Number analyzed (Participants) | 188 | 190
percentage of patients
  Day 5: Composite Cure | 89.4 | 94.2
  Day 5: Composite Failure | 10.6 | 5.8

4. Secondary Outcome: Percentage of Patients With Composite of Microbiological Eradication and Clinical Cure in the ME Population at TOC
Description: Microbiological eradication: urine culture showed the pathogen found at baseline at ≥10^5 CFU/mL was reduced to <10^4 CFU/mL. Clinical Cure TOC: Complete resolution or return to premorbid levels of core symptoms of cUTI and no new symptoms develop, and no use of non-study antibiotic therapy for the current cUTI. Failure TOC: Persistence of one or more core symptom of infection or reappearance of or development of new core symptoms that require alternative non-study antibiotic therapy for the current cUTI.
Time Frame: Day 17 TOC Visit
Population: The ME (TOC) population consists of clinically evaluable patients with interpretable culture results at TOC, defined as one that has clearly identified pathogen(s) or one where baseline pathogen(s) could be excluded.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin | Meropenem
Number analyzed (Participants) | 179 | 177
percentage of patients
  TOC: Composite Cure | 84.9 | 75.1
  TOC: Composite Failure | 15.1 | 24.9

5. Secondary Outcome: Percentage of Patients With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence associated with the use of a drug in humans, whether or not it is considered to be drug related. An AE (also referred to as an adverse experience) can be any unfavorable and unintended sign (eg, an abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, and it does not imply any judgment about causality. Adverse events also include the exacerbation or worsening of a condition present at screening other than the index infection for which the patient was enrolled in the study. A TEAE is any AE that newly appeared, increased in frequency, or worsened in severity following initiation of study drug.
Time Frame: Up to Day 32
Population: The safety population included all randomized patients who received any amount of study drug.
Measure: Number; unit: percentage of patients
Arm/Group | Plazomicin | Meropenem
Number analyzed (Participants) | 303 | 301
percentage of patients | 19.5 | 21.6

6. Secondary Outcome: Plasma Pharmacokinetics (PK): Area Under the Curve From 0 to 24 Hours (AUC 0-24h)
Description: PK blood samples were collected on Day 3 (plus or minus 1 day) of study drug administration for the determination of plazomicin concentrations in plazomicin-treated patients.
Time Frame: Day 3
Population: The PK Population included patients who received at least one dose of plazomicin and had at least one quantifiable plazomicin plasma concentration available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*h/L (milligrams times hour per liter)
Arm/Group | Plazomicin
Number analyzed (Participants) | 281
mg*h/L (milligrams times hour per liter) | 234 (38.5)

7. Secondary Outcome: Plasma PK: Maximum Observed Plasma Drug Concentration (Cmax)
Description: as for outcome 6
Time Frame: Day 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Plazomicin
Number analyzed (Participants) | 281
mg/L | 46.6 (43)

8. Secondary Outcome: Plasma PK: Minimum Observed Plasma Drug Concentration (Cmin)
Description: as for outcome 6
Time Frame: Day 3
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Plazomicin
Number analyzed (Participants) | 281
mg/L | 0.88 (95.4)

ADVERSE EVENTS:
Time Frame: Up to Day 32
Description: The AE collection period began with the first dose of study drug and ended at the last follow up visit (LFU). LFU was up to 32 Days after the first dose of study drug.
Arm/Group | Plazomicin | Meropenem
All-Cause Mortality (participants affected / at risk) | 1/303 | 0/301
Serious Adverse Events (participants affected / at risk) | 5/303 | 5/301
Other Adverse Events (participants affected / at risk) | 0/303 | 0/301
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Plazomicin (N=303) | Meropenem (N=301)
Metastatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 0 | 1
Orchitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 0 | 1
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Investigator may publish/present the study results provided all of the following: (i) the primary publication has been published; or, if no such publication has occurred, at least 18m have passed since the completion of the study; (ii) Achaogen is allowed at least 60d to review; (iii) confidential information is deleted as requested; (iv) comments and proposed revisions are considered; and (v) during the 60d review, if requested, the Investigator shall delay the publication or presentation.